CLINICAL TRIAL: NCT03973554
Title: Caries Prevention Potential of Pearl Powder Versus Casein Phosphopeptide-amorphous Calcium Phosphate on Enamel White Spot Lesions: Randomized Clinical Trial.
Brief Title: Caries Prevention Potential of Pearl Powder Versus CPP-ACP on Enamel White Spot Lesions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruba Alaa El Din Adel El Damarisy (Other)
Responsible Party: Sponsor-Investigator, Ruba Alaa El Din Adel El Damarisy, principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11090
Record Dates: First submitted 2019-06-01; First posted 2019-06-04 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: White Spot Lesion of Tooth
Keywords: white spot lesions,; pearl powder; CPP-ACP
MeSH Terms: interventions — pearl powder; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pearl powder (Experimental): natural product, support bone and joint health
  Interventions: Other: pearl powder
- CPP-ACP (Active Comparator): product for professional use containing the active ingredient (CPP-ACP), a special milk-derived protein that has a unique ability to release bio-available calcium and phosphate to tooth surfaces.
  Interventions: Drug: CPP-ACP

INTERVENTIONS:
Other: pearl powder — natural product, support bone and joint health
  Arms: pearl powder
Drug: CPP-ACP — Remineralising sugar free dental topical crème, containing bio-available calcium and phosphate
  Other Names: tooth mousse
  Arms: CPP-ACP

SUMMARY:
to evaluate the caries prevention potential of pearl powder against CPP-ACP in enamel white spot lesions.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the caries prevention potential of pearl powder against CPP-ACP in enamel White Spot Lesions using laser fluorescence device scoring from 0 to 99, with daily application time of 3 months and follow up period of 6,9,and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* good oral hygiene
* cooperative patient
* completion of orthodontic therapy
* presence of at least two white spot lesions on the labial surface of six maxillary anterior teeth, that were not present before orthodontic treatment

Exclusion Criteria:

* bad oral hygiene
* lack of patients compliance
* allergy to milk products
* pregnant or lactating women
* presence of dentin caries, restorations, or enamel hypoplasia on maxillary anterior teeth
* presence of periodontal pockets around maxillary anterior teeth

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-10-30 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
caries prevention in enamel white spot lesion | 12 months
  caries prevention using laser fluorescence device

CONTACTS AND LOCATIONS:
Overall Officials: Ruba A El Damarisy, MDS, Principal Investigator — Cairo University